CLINICAL TRIAL: NCT04025723
Title: Differences in Rate of Recovery Between Young and Middle-aged Men After Downhill Running
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Gepner Yftach (Other)
Responsible Party: Sponsor-Investigator, Gepner Yftach, Principal Investigator, Tel Aviv University
Organization: Tel Aviv University (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: Recovery
Record Dates: First submitted 2019-07-09; First posted 2019-07-19 (Actual); Last update posted 2021-03-25 (Actual); Status verified 2021-03

CONDITIONS: Exercise
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Intervention Model Description: Young (18-30 y) and middle aged (35-50 y) men will perform 60 min of downhill running
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Young (Active Comparator): men aged between 18 to 30 years old
  Interventions: Other: Downhill running
- Middle-aged (Active Comparator): men aged between 35 to 50 years old
  Interventions: Other: Downhill running

INTERVENTIONS:
Other: Downhill running — 60 minutes downhill running in 10% grade, in an effort of 65% of VO2max.

SUMMARY:
The aim of this study is to evaluate differences in rate of recovery between young and middle-aged men after prolonged (downhill) running. Thirty healthy young (n=15, 18-30 y) and middle-aged (n=15, 35-50y) men will be recruited for this study. Participants will perform 60 minutes of downhill run at 65% of their maximal oxygen consumption (VO2max). Recovery parameters will be evaluated during 48 hours following the downhill protocol, and will include changes in performance tests, inflammatory markers, muscle integrity and heart-rate variability. Questioners will be used to evaluate muscle soreness and fatigue. We hypothesized that middle-aged males will have longer rate of recovery following the downhill running protocol, as compared to younger age males.

ELIGIBILITY:
Inclusion Criteria:

* Active man which perform a minimum of 150 minutes/week of exercise
* Able to complete 60 min run.

Exclusion Criteria:

* Injuries in lower body
* cardio-respiratory disease
* supplementing with performance enhancing supplements

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2020-02-20 (Actual); Primary Completion 2021-01-16 (Actual); Study Completion 2021-01-16 (Actual)

PRIMARY OUTCOMES:
Changes over time in Maximal voluntary contraction (MVC) of the Musculus quadriceps femoris | MVC will be measured before and after 30, 60, 120 minutes (Day 0), 24 (Day 1) and 48 hours (Day 2) after the downhill running
  MVC (kg) measures the greatest amount of tension a muscle can generate and hold. We will measure it before (baseline) and after the downhill running protocol. Changes from baseline will be calculated for each time point. A comparison of the changes in MVC over time will be made between the two study's arms .
Changes over time in vertical jump (VJ) | VJ will be measured before and after 30, 60, 120 minutes (Day 0), 24 (Day 1) and 48 hours (Day 2) after the downhill running
  VJ (cm) is the height achieved after a vertical jump.We will measure it before (baseline) and after the downhill running protocol. Changes from baseline will be calculated for each time point. A comparison of the changes in VJ over time will be made between the two study's arms .
Changes over time in stride length | Stride length will be measured before and after 30, 60, 120 minutes (Day 0), 24 (Day 1) and 48 hours (Day 2) after the downhill running
  Stride length (cm) is the distance achieved while walking or running and is calculated as the distance from the toe of your right foot (starting position) to the toe of your right foot (ending position). Participants will run on a treadmill with pressure sensors for 2 minutes. We will measure stride length before (baseline) and after the downhill running protocol. Changes from baseline will be calculated for each time point. A comparison of the changes in stride length over time will be made between the two study's arms .
Changes over time in stride frequency | Stride frequency will be measured before and after 30, 60, 120 minutes (Day 0), 24 (Day 1) and 48 hours (Day 2) after the downhill running
  Stride frequency (strides per minutes) is the number of times a single foot hits the ground while walking or running. Participants will run on a treadmill with pressure sensors for 2 minutes. We will measure stride frequency before (baseline) and after the downhill running protocol. Changes from baseline will be calculated for each time point. A comparison of the changes in stride frequency over time will be made between the two study's arms .

SECONDARY OUTCOMES:
Changes over time in the concentration of circulating interleukin -6 (IL-6) | The circulating parameters will be measured before and after 30, 60, 120 minutes (Day 0), 24 (Day 1) and 48 hours (Day 2) after the downhill running
  Concentration of circulating IL-6 (pg/ml) will be measured before (baseline) and after the downhill running protocol. Changes from baseline will be calculated for each time point. A comparison of the changes in concentration of circulating IL-6 over time will be made between the two study's arms .
Changes over time in the concentration of circulating interleukin -10 (IL-10) | The circulating parameters will be measured before and after 30, 60, 120 minutes (Day 0), 24 (Day 1) and 48 hours (Day 2) after the downhill running
  Concentration of circulating IL-10 (pg/ml) will be measured before (baseline) and after the downhill running protocol. Changes from baseline will be calculated for each time point. A comparison of the changes in concentration of circulating IL-6 over time will be made between the two study's arms .
Changes over time in the concentration of circulating interleukin -1 receptor antagonist (IL-1ra) | The circulating parameters will be measured before and after 30, 60, 120 minutes (Day 0), 24 (Day 1) and 48 hours (Day 2) after the downhill running
  Concentration of circulating IL-1ra (pg/ml) will be measured before (baseline) and after the downhill running protocol. Changes from baseline will be calculated for each time point. A comparison of the changes in concentration of circulating IL-6 over time will be made between the two study's arms .
Changes over time in the concentration of circulating tumor necrosis factor alpha (TNFa) | The circulating parameters will be measured before and after 30, 60, 120 minutes (Day 0), 24 (Day 1) and 48 hours (Day 2) after the downhill running
  Concentration of circulating TNFa (pg/ml) will be measured before (baseline) and after the downhill running protocol. Changes from baseline will be calculated for each time point. A comparison of the changes in concentration of circulating IL-6 over time will be made between the two study's arms .
Changes over time in the concentration of circulating c-reactive protein (CRP) | The circulating parameters will be measured before and after 30, 60, 120 minutes (Day 0), 24 (Day 1) and 48 hours (Day 2) after the downhill running
  Concentration of circulating CRP (nmol/L) will be measured before (baseline) and after the downhill running protocol. Changes from baseline will be calculated for each time point. A comparison of the changes in concentration of circulating IL-6 over time will be made between the two study's arms .
Changes over time in the concentration of circulating creatine kinase (CK) | The circulating parameters will be measured before and after 30, 60, 120 minutes (Day 0), 24 (Day 1) and 48 hours (Day 2) after the downhill running
  Concentration of circulating CK (IU/L) will be measured before (baseline) and after the downhill running protocol. Changes from baseline will be calculated for each time point. A comparison of the changes in concentration of circulating IL-6 over time will be made between the two study's arms .
Changes over time in the concentration of circulating lactate dehydrogenase (LDH) | The circulating parameters will be measured before intervention, immediately after, 30, 60, 120 minutes, 24 and 48 h post intervention.
  Concentration of circulating LDH (IU/L) will be measured before (baseline) and after the downhill running protocol. Changes from baseline will be calculated for each time point. A comparison of the changes in concentration of circulating IL-6 over time will be made between the two study's arms .
Changes over time in muscle fibers morphology | MRI will be conducted up to 1 week before the intervention (screening day, Day -1) and after 24 hours (Day 1) or 48 hours (Day 2) post downhill running.
  Muscle fibers morphology of the Musculus quadriceps femoris will be assessed by Diffusion Tensor Imaging by magnetic resonance imaging (MRI). We will assess muscle fiber morphology before (baseline) and 48 hours after the downhill running protocol. Changes from baseline will be calculated for each time point. A comparison of the changes in muscle fiber morphology over time will be made between the two study's arms .
Changes over time in delayed-onset muscle soreness (DOMS) | DOMS will be measured before intervention, immediately after, 30, 60, 120 minutes after (Day 0), 24 hours (Day 1) and 48 hours (Day 2) post downhill running.
  DOMS will be evaluated using the Visual Analogue Scale (VAS). The VAS scale will be 150 mm line with "no pain" on one side and "maximal pain" on the other. Each participant will mark a line based on his soreness in the Musculus quadriceps femoris and Musculus gastrocnemius. The distance (mm) from the "no pain" side will be measured. DOMS assessment will be made before (baseline) and after the downhill running protocol. Changes from baseline will be calculated for each time point.
Changes over time in Mood States | Changes in Mood States will be measured before intervention, immediately after, 30, 60, 120 minutes after (Day 0), 24 hours (Day 1) and 48 hours (Day 2) post downhill running.
  Changes in mood state will be assessed using the Profile of Mood States questioner (POMS). POMS is a validated questioners comprised from 58 feelings and emotions. For each parameter, the participants will be asked how he feels right know and select a value ranging between 0 to 4, where "0" means "not at all" and "4" means "extremely". A Total Mood Disturbance (TMD) score is calculated by summing the totals for the negative sub-scales and then subtracting the totals for the positive sub-scales.
Changes over time in total fatigue | Changes in total fatigue will be measured before intervention, immediately after, 30, 60, 120 minutes after (Day 0), 24 hours (Day 1) and 48 hours (Day 2) post downhill running.
  Changes in total fatigue will be assessed using the Rating Of Fatigue scale (ROF). ROF is a validated 11-point numerical scale ranging from zero to ten. Participants will be asked to rate how fatigued they feel whereas, "0" is "not fatigued at all" and "10" is "Total fatigue and exhaustion- nothing left". Total fatigue assessment will be made before (baseline) and after the downhill running protocol. Changes from baseline will be calculated for each time point.
Changes over time in none-specific muscle fatigue- MVC of the forearm | None-specific muscle fatigue tests will be measured before intervention, immediately after, 30, 60, 120 minutes after (Day 0), 24 hours (Day 1) and 48 hours (Day 2) post downhill running.
  We will measure none-specific muscle fatigue using hand gripper to evaluate the forearm MVC (kg). We will measure it before (baseline) and after the downhill running protocol. Changes from baseline will be calculated for each time point. A comparison of the changes in MVC over time will be made between the two study's arms .
Changes over time in heart rate variability (HRV) | Between 3 to 5 days before screening day (Day -1) and downhill running (Day 0) for baseline assessment, and after the downhill running (Day 0) until day 2
  HRV (ms) quantifies the variability between heart beats. We will use the time-based analysis and the root mean square of successive differences of R-R intervals (RMSSD) value. The measurements will be done continuously with a heart rate monitor. Baseline measurements will be done for 3 to 5 days before the downhill running and the average value will be defined as "baseline HRV". Changes in HRV will be measured continuously in the 48 hours following the running. Percentage from "baseline HRV" will be calculated and compared between the two study's arms.

CONTACTS AND LOCATIONS:
Locations (1):
- Tel Aviv University, Tel Aviv, Israel